CLINICAL TRIAL: NCT00744874
Title: Multi-Array Ablation of the Pulmonary Veins for Paroxysmal Atrial Fibrillation
Brief Title: Ablation of the Pulmonary Veins for Paroxysmal Afib
Acronym: MAP-PAF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFI-40
Record Dates: First submitted 2008-08-28; First posted 2008-09-01 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ablated Patients (Experimental): Patients with a history of symptomatic paroxysmal (self-terminating) AF and meeting all inclusion/exclusion criteria, as identified by the clinical investigator, will be enrolled in the study.
  Interventions: Procedure: RF Ablation procedure

INTERVENTIONS:
Procedure: RF Ablation procedure — Patients with a history of symptomatic paroxysmal (self-terminating) AF and meeting all inclusion/exclusion criteria, as identified by the clinical investigator, will be enrolled in the study.
  Other Names: Radio Frequency Ablation

SUMMARY:
The purpose of this trial was to investigate and confirm the safety, efficacy, and efficiency of the Ablation Frontiers® Cardiac Ablation System when used in the treatment of paroxysmal atrial fibrillation. (PAF)

DETAILED DESCRIPTION:
This trial was a non-randomized, multi-center, prospective study of subjects with symptomatic, paroxysmal atrial fibrillation (PAF). The purpose of this study was to investigate and confirm the safety, efficacy and efficiency of the Medtronic Ablation Frontiers® Cardiac Ablation System when used for the treatment of paroxysmal AF. The trial was conducted over a 2 year period with enrollment occurring between 4 October 2007 and 1 December 2008.

ELIGIBILITY:
Inclusion Criteria:

History of symptomatic paroxysmal atrial fibrillation defined as:

* Self terminating AF lasting no more than 7 days
* AF events demostrating spontaneous conversion back to sinus rhythm
* Documentation of one or more events with PAF tracings by ECG, event recordings, pacemaker strips or monitor rhythm strips within the past year
* AF symptoms defined as the manisfestation of any of the following: Palpitations, Fatigue, Exertional dyspnea, effort intolerance
* Age between 18 and 70
* Willingness, ability and commitment to participate in baseline and follow-up evaluations for the full length of the study

Exclusion Criteria:

* Structural heart disease of clinical significance
* Prior ablation for arrhythmias other than AF within the past three months
* Prior left sided AF ablation
* Enrollment in any other ongoing arrhythmia study protocol
* Any ventricular tachyarrhythmias currently being treated where the arrhythmia or the management may interfere with this study
* Active infection or sepsis
* Any history of cerebral vascular disease including stroke or TIAs
* Pregnancy or lactation
* Untreatable allergy to contrast media
* Any diagnosis of atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or any other reversible or non-cardiovascular causes
* History of blood clotting (bleeding or thrombotic) abnormalities
* Known sensitivities to heparin or warfarin
* Severe COPD (identified by an FEV1 < 1)
* Severe co morbidity or poor general physical/mental health that, in the opinion of the investigator, will not allow the patient to be a good study candidate (i.e. other disease processes, mental capacity, substance abuse, shortened life expectance, etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-10; Primary Completion 2009-09 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Hjertecenter Varde, Varde
- Zentralklinik, Bad Berka, Germany
- St. Antonius Ziekenhuis, Nieuwegein, Netherlands
- Klinik im Park, Zurich, Switzerland

REFERENCES:
- See also: Company website — http://www.ablationfrontiers.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Ablated Participants: Participants that who had a pulmonary vein isolation procedure performed with the Medtronic Ablation Frontiers® Cardiac Ablation System for the treatment of atrial fibrillation.
Period: Overall Study
Arm/Group | Ablated Participants
Started | 55
Completed | 51
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Not completed — Study Device not available at procedure | 1
Not completed — Unable to accomodate schedule | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ablated Participants
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 34
Region of Enrollment [Number; unit: participants]
  Denmark | 18
  Germany | 7
  Netherlands | 21
  Switzerland | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Pulmonary Vein Isolation
Description: Acute effectiveness was defined as successful isolation of all pulmonary veins. Pulmonary vein isolation was documented by the absence of pulmonary vein potentials when assessed by electrogram tracings in sinus rhythm using the PVAC catheter.
Time Frame: 6 months
Population: Subjects that had successful pulmonary vein isolation.
Measure: Number; unit: participants
Arm/Group | Ablated Participants
Number analyzed (Participants) | 55
participants | 53

2. Primary Outcome: Chronic Effectiveness
Description: The primary endpoint for chronic effectiveness was the evaluation of the proportion of subjects with treatment success computed at the 6 month visit. In order to be classified as a chronic success, all subjects were required to meet the following criteria: Absence of clinically significant AF (greater than 60 seconds) or left atrial tachycardia recorded on a 7-day Holter, absence of symptomatic AF after a 3 month blanking period, off all Class I and III AADs at 6 months.
Time Frame: 6 months
Population: The primary endpoint for chronic effectiveness was the evaluation of the proportion of subjects with treatment success computed at the 6 month visit.
Measure: Number; unit: participants
Arm/Group | Ablated Participants
Number analyzed (Participants) | 55
participants | 10 [9.1 to 30.9]

3. Primary Outcome: Acute Safety
Description: The Acute Safety Endpoint was defined as the proportion of subjects with Serious Adverse Events (SAEs) that were procedure- and/or device-related within 7 days after the ablation procedure. The relatedness of each event was assessed by the investigator at each site.
Time Frame: 7 days post procedure
Population: The proportion of subjects with one or more serious procedure and/or device related AEs occurring within 7 days of the ablation procedure. No acute events were related to the device.
Measure: Number; unit: participants
Arm/Group | Ablated Participants
Number analyzed (Participants) | 55
participants | 2

4. Primary Outcome: Chronic Safety
Description: The Chronic Safety Endpoint was the proportion of subjects with serious procedure- and/or device-related events in the 7 day to 6 month follow-up period post-ablation. The relatedness of each event was assessed by the investigator at each site.
Time Frame: 7 day post procedure to 6 months
Population: The Chronic Safety Endpoint is the proportion of subjects with serious procedure and/or device-related events in the 7 day to 6 month follow-up period post-ablation. The relatedness of each event was assessed by the investigator at each site.
Measure: Number; unit: participants
Arm/Group | Ablated Participants
Number analyzed (Participants) | 55
participants | 0

5. Secondary Outcome: Atrial Fibrillation Symptom Severity Scores From Baseline to 6 Months
Description: Subjects rated the severity of their AF-related symptoms at baseline and at each follow-up visit for the study. Symptoms that were assessed at each visit included the presence of palpitations, fatigue, shortness of breath, lightheadedness or dizziness, and/or lack of energy upon exertion or exercise. Each symptom was rated on a scale from 1 (no symptoms) to 5 (most severe). Total scores were obtained by adding up the rating for each symptom to obtain a range of results between 5 (asymptomatic) to 25 (severely symptomatic).
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ablated Patients Symptom Severity Score at Baseline: Participants that who had a pulmonary vein isolation procedure performed with the Medtronic Ablation Frontiers® Cardiac Ablation System for the treatment of atrial fibrillation.Measured scores at baseline.
- Ablated Patients Symptom Severity Score at 3 Months: Participants that who had a pulmonary vein isolation procedure performed with the Medtronic Ablation Frontiers® Cardiac Ablation System for the treatment of atrial fibrillation.Measured scores at 3 months after the procedure.
- Ablated Patients Symptom Severity Score at 6 Months: Participants that who had a pulmonary vein isolation procedure performed with the Medtronic Ablation Frontiers® Cardiac Ablation System for the treatment of atrial fibrillation.Measured scores at 6 months after the procedure.
Arm/Group | Ablated Patients Symptom Severity Score at Baseline | Ablated Patients Symptom Severity Score at 3 Months | Ablated Patients Symptom Severity Score at 6 Months
Number analyzed (Participants) | 54 | 50 | 51
units on a scale
  Palpitations | 3.4 (1) | 1.9 (1) | 1.9 (1)
  Fatigue | 3.2 (1.1) | 2 (1.2) | 1.9 (1.1)
  Shortness of Breath | 2.7 (1.2) | 1.9 (1.1) | 1.8 (1.1)
  Lightheadedness / Dizziness | 2.7 (1.2) | 1.5 (0.9) | 1.5 (1)
  Lack of Energy During Exertion or Exercise | 3.3 (0.9) | 2.1 (1.1) | 2.1 (1.3)
  Total AF Symptom Severity Score | 15.4 (4.1) | 9.4 (4.4) | 9.2 (4.7)

6. Secondary Outcome: The Short Form 36 Question (SF-36) Health Survey Quality of Life Survey at 6 Months Compared to Baseline
Description: The SF-36 is a short-form health survey of 36 questions that yields an 8-scale health profile as well as psychometrically-based physical and mental health summary measures. In order to assess improvement in self-perceived quality of life, subjects were asked to complete SF-36 questionnaires at baseline and at each follow-up visit. The results of the Physical Component and Mental Component scores from the two summary measures that aggregate sub-scales were then compared.The SF-36 subscales range from 0 (lowest) to 100 (highest). The subscales are averaged together for a total score between 0 to 100. A higher score represents a better outcome when compared to a lower score.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline Quality of Life Scores: Quality of life scores at baseline or before pulmonary vein isolation procedure was performed with the Medtronic Ablation Frontiers® Cardiac Ablation System for the treatment of atrial fibrillation.
- Quality of Life Scores at 3 Months: Quality of life scores at 3 months or 3 months before pulmonary vein isolation procedure was performed with the Medtronic Ablation Frontiers® Cardiac Ablation System for the treatment of atrial fibrillation.
- Quality of Life Scores at 6 Months: Quality of life scores at 6 months or 6 months before pulmonary vein isolation procedure was performed with the Medtronic Ablation Frontiers® Cardiac Ablation System for the treatment of atrial fibrillation.
Arm/Group | Baseline Quality of Life Scores | Quality of Life Scores at 3 Months | Quality of Life Scores at 6 Months
Number analyzed (Participants) | 48 | 50 | 51
units on a scale
  Physical Component Score | 46.4 (9.7) | 50.4 (9.2) | 51.8 (8.1)
  Mental Compnent Score | 46.8 (11.7) | 49.4 (10) | 51.6 (9)

7. Secondary Outcome: Measurement of the Cumulative RF Time for Pulmonary Vein(PV)Isolation of All Accessible Pulmonary Veins
Description: Cumulative RF time was calculated by the difference between the start time of catheter ablations and the end time of the ablation
Time Frame: After Procedure
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Cumulative Radio Frequency Time for PV Isolation: Participants that who had a pulmonary vein isolation procedure performed with the Medtronic Ablation Frontiers® Cardiac Ablation System for the treatment of atrial fibrillation.
Arm/Group | Cumulative Radio Frequency Time for PV Isolation
Number analyzed (Participants) | 53
minutes | 56.3 (37.1)

8. Secondary Outcome: Total Procedure Time
Description: Measurement of total procedure time defined as "skin to skin" and left atrial dwell time (transseptal puncture to removal of all left atrial catheters)
Time Frame: End of Procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ablated Participants
Number analyzed (Participants) | 54
minutes | 117.9 (58.2)

9. Secondary Outcome: Total Fluoroscopy Time
Description: Total time that flouroscopy was used during the ablation procedure.
Time Frame: Post Ablation Procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ablated Participants
Number analyzed (Participants) | 53
minutes | 26 (15.4)

ADVERSE EVENTS:
Time Frame: All adverse events were collected up to 6 months.
Description: The seriousness and relatedness of all AEs were assessed by the investigator at each site. The AE's included: Cerobrovascular accident, Major bleeding, Cardiac tamponade, Pulmonary vein stenosis, Pericarditis, Myocardial infarction, Diaphragmatic paralysis, Atrio-esophageal fistula, and Death.
Arm/Group | Ablated Participants
Serious Adverse Events (participants affected / at risk) | 9/55
Other Adverse Events (participants affected / at risk) | 19/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ablated Participants (N=55)
Bleeding (Surgical and medical procedures) | 1 (1)
Chest Discomfort (Surgical and medical procedures) | 1 (1)
Collapse After AF recurrence (Cardiac disorders) | 1 (1)
Arrythmia, pro arrhythmia (Cardiac disorders) | 3 (3)
Dizziness (General disorders) | 1 (1)
Sudden Deafness followed by tinnitus (Ear and labyrinth disorders) | 1 (1)
Heart Catheterization (Surgical and medical procedures) | 1 (1)
Cerebrovascular Accident- Ischemic attack (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ablated Participants (N=55)
Back pain (General disorders) | 1 (1) — Back pain as a result of a car accident
Arrythmia, proarrythmia (Cardiac disorders) | 14 (16)
Fatigue (General disorders) | 1 (1)
Headache (General disorders) | 2 (2) — Headache as a result of a car accident.
Allergic reaction (Immune system disorders) | 1 (1) — Allergic reaction to contrast media.
Dizziness (General disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 3 (3)
Cerebrovascular Accident/ Ischemic Attack (Vascular disorders) | 1 (1)
Infections (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less